CLINICAL TRIAL: NCT00244881
Title: A Phase II Study of AZD2171 in Breast Cancer Stage IV (10006202)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02937; 05-160; U01CA062490 (NIH); CDR0000445438 (Registry Identifier: PDQ (Physician Data Query)); NCT00215488 (obsolete NCT alias)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2013-11

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — cediranib

ARMS (1):
- Treatment (cediranib maleate) (Experimental): Patients receive oral AZD2171 once daily for 42 days. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cediranib maleate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: AZD2171; Recentin
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
AZD2171 (cediranib maleate) may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. This phase II trial is studying how well AZD2171 works in treating patients with refractory stage IV breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluation of the fraction of patients with increased levels of circulating endothelial cells after 3 weeks of treatment with AZD2171.

II. Estimation of the objective response rate (ORR = CR + PR) among patients with refractory breast cancer receiving AZD2171.

SECONDARY OBJECTIVES:

I. Estimation of the response/stable disease rate (RSDR = CR + PR + SD). II. Characterization of the toxicity associated with AZD2171 in this cohort of patients.

III. Analyses to correlate serial quantification of circulating endothelial cells and circulating tumor cells with traditional clinical endpoints including RR and TTP.

IV. Develop pharmacodynamic measures of AZ2171 activity based on monocyte count and VEGFR-1 phosphorylation within monocytes.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive oral AZD2171 once daily for 42 days. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 3 months.

PROJECTED ACCRUAL: A total of 26 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed Breast Cancer, stage IV, including:

  * "Breast neoplasms malignant and unspecified (incl nipple)","Breast and nipple neoplasms malignant","Breast cancer stage IV","10006202"
  * Breast neoplasms malignant and unspecified (incl nipple)","Breast and nipple neoplasms malignant","Breast cancer recurrent","10006198"
  * "Breast neoplasms malignant and unspecified (incl nipple)","Breast and nipple neoplasms malignant","Inflammatory carcinoma of breast stage IV","10021979"
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Patients must have refractory breast cancer, defined as overt clinical tumor progression on most recent treatment with either hormonal therapy, chemotherapy, and/or trastuzumab therapy; patients with up to 3 prior chemotherapy regimens and with any number of biological (hormonal, trastuzumab) regimens for metastatic breast cancer will be eligible
* Life expectancy of greater than 3 months as assessed by the patient's primary oncologist
* Absolute neutrophil count > 1,500/mcL
* Platelets > 100,000/mcL
* Hemoglobin >= 8 g/dL
* Prothrombin time < institutional upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN
* AST(SGOT)/ALT(SGPT) =< 2.5 × ULN
* Creatinine within normal institutional limits
* Urinalysis with < 1+ proteinuria
* Troponin T or I within normal institutional limits
* LVEF >= 45%, as assessed by echocardiogram or nuclear medicine gated study, within 30 days prior to initiating protocol-based treatment
* At present, the potential of AZD2171 for clinically significant drug interactions involving the CYP isozymes is unknown; however, studies of the agent in rats indicated possible suppression of CYP1A that may be of biological significance; eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or PK of AZD2171 will be determined following review of their case by the Principal Investigator.
* AZD2171 has been shown to terminate fetal development in the rat, as expected for a process dependent on VEGF signaling; for this reason, women of child-bearing potential must have a negative pregnancy test prior to study entry; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* No therapeutic anti-coagulation; the use of low dose warfarin (1-2 mg/day), intermittent doses of TPA (2 mg x 1), or heparin flushes to prophylax against central venous catheter-associated clots is acceptable
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy, or major surgery within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents nor have participated in an investigational trial within the past 30 days
* Patients may not have been previously treated with an anti-angiogenesis agent
* \Patients may not be receiving any medication that may markedly affect renal function (e.g., vancomycin, amphotericin, pentamidine); these medications will also not be permitted after the start of the study
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; a head CT or MRI must be performed at baseline
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD2171
* Any contraindications/barrier to oral medication
* EKG abnormalities of known clinical significance, such as prolonged QT (mean QTc > 470 msec, with Bazett's correction, in screening electrocardiogram or history of familial long QT syndrome); an EKG is required for study entry
* Uncontrolled intercurrent illness including, but not limited to hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because AZD2171 is a VEGF inhibitor with known abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD2171, breastfeeding should be discontinued if the mother is treated with AZD2171
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD2171; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients at increased risk for compromised LVEF requiring concurrent use of drugs or biologics with proarrythmic potential; these drugs are prohibited during studies with AZD2171 (refer to Appendix J for a listing of these agents)
* Patients with a New York Heart Association classification of III or IV are excluded (NOTE: patients classified as class II are eligible if controlled on medication and stable with increased monitoring)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-09; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold Burstein, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Dana-Farber/Harvard Cancer Center
Period: Overall Study
Arm/Group | Treatment (Cediranib Maleate)
Started | 26
Completed | 23
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Fraction of Patients With Increased Levels of Circulating Endothelial Cells
Description: An exact 95% confidence interval (CI) will be calculated for the CEC response rate. With 26 patients, this CI will be no wider than 40% (e.g., if 13 of 26 patients respond, the CI is 30% to 70%).
Time Frame: After 3 weeks of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 26
percentage of participants | 30

2. Primary Outcome: Objective Response Rate (ORR = CR + PR) Classified According to RECIST Criteria
Description: RECIST 1.0 Criteria
Time Frame: Up to 7 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 26
percentage of participants | 8 [1 to 25]

3. Secondary Outcome: Response/Stable Disease Rate Defined as the Percentage of Patients Demonstrating CR + PR + SD
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Cediranib Maleate)
Number analyzed (Participants) | 26
percentage of participants | 45

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment (Cediranib Maleate)
Serious Adverse Events (participants affected / at risk) | 7/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cediranib Maleate) (N=26)
Vomiting (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 (1)
Gallbladder Abnormality (Gastrointestinal disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cediranib Maleate) (N=26)
Hypertension (Cardiac disorders) | 21 (21)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Fatigue (General disorders) | 10 (10)
Proteinuria (Renal and urinary disorders) | 8 (8)
Esophagitis/Mucositis (Gastrointestinal disorders) | 7 (7)
LFT Abnormalities (Cardiac disorders) | 7 (7)
Hypothyroidism (Endocrine disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
LV systolic dysfunction (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less